CLINICAL TRIAL: NCT06348381
Title: Prediction of Anastomotic Complications and Recurrent Laryngeal Nerve Injury Based on Postoperative Early Endoscopic Evaluation: a Prospective, Observational, Non-interventional Study
Brief Title: Prediction of Anastomotic Complications and Recurrent Laryngeal Nerve Injury Based on Postoperative Early Endoscopic Evaluation
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Li, Deputy director of department of thoracic surgery, Shanghai Chest Hospital
Other Study IDs: IS24030
Record Dates: First submitted 2024-03-30; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Neoplasm; Anastomotic Leak; Recurrent Laryngeal Nerve Injuries; Anastomotic Stenosis; Endoscopic Evaluation
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak; Recurrent Laryngeal Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Analyze the correlation between the conformity of the anatomy (based on endoscopic examination) and postoperative anastomotic fistula and anastomotic stenosis; establish an anastomotic classification; and construct a predictive model combined with perioperative-related test indicators to provide more accurate risk assessment for clinical practice. Analyze the natural recovery process of postoperative recurrent laryngeal nerve injury in esophageal cancer by tracking vocal cord movement (based on endoscopic examination) and hoarseness symptoms; combined with perioperative related surgical and laboratory indicators, identify the relevant risk factors associated with delayed recovery of recurrent laryngeal nerve injury.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with esophageal squamous cell carcinoma;
2. 18 - 80 years old;
3. ECOG PS 0-1;
4. Thoracic esophageal cancer (20-40cm from the incisors);
5. Received radical resection of esophageal cancer in our hospital from April 2024 to July 2024;
6. Received the McKeown procedure in our hospital's single treatment group;
7. Received gastric reconstruction and cervical anastomosis with a side-to-side anastomotic device;
8. Complete clinical materials.

Exclusion Criteria:

1. History of other malignant tumors;
2. Incomplete or missing clinical materials;
3. Received combined surgery (total laryngectomy + esophagectomy, esophagectomy + lung resection, esophagectomy + aorta, etc.);
4. Gastric reconstruction or cervical anastomosis with a side-to-side anastomotic device was not performed;
5. Patients who underwent 3-field lymph node dissection;
6. Patients with clear intraoperative recurrent laryngeal nerve section;
7. Highly suspected anastomotic fistula before the first endoscopic evaluation (abnormal secretion at the cervical anastomotic site, abnormal drainage fluid in the chest tube, and high fever that other reasons cannot explain);
8. Lost to follow-up.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who received radical resection of esophageal cancer in our hospital from April 2024 to July 2024.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak | One week to six months after esophagectomy
  leak of the anastomosis
anastomotic stenosis | One week to six months after esophagectomy
  stenosis of anastomosis
laryngeal nerve injury | One week to six months after esophagectomy
  hoarseness symptoms, recovery progression of recurrent laryngeal nerve injury

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided